CLINICAL TRIAL: NCT06859359
Title: Improving Maternal Cardiovascular Outcomes Through the Implementation of a Hypertensive Disorders of Pregnancy Bundle in Nigeria
Acronym: IMPACT-HDP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Zainab Mahmoud, Assistant Professor of Medicine, Washington University School of Medicine
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 202311185; K23HL173684 (NIH)
Record Dates: First submitted 2024-11-06; First posted 2025-03-05 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-02

CONDITIONS: Hypertensive Disorder of Pregnancy
Keywords: Hypertension; Pregnancy; Preeclampsia; HDP
MeSH Terms: conditions — Toxemia; Hypertension; Pre-Eclampsia

STUDY DESIGN:
Intervention Model Description: Type 1 hybrid stepped-wedge cluster randomized trial to assess if the utilization of the HDP Implementation Bundle will improve postpartum BP among women with HDP in Nigeria. Randomization will be done at cluster level and sites will begin in control and cross over to intervention phase
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Phase: For capturing baseline parameters. (No Intervention): In the control phase, baseline data including postpartum BP measurement, treatment at enrollment and BP at 6- and 12-weeks follow-up will be recorded. BP control rates, and clinical outcomes will also be recorded.
- Intervention Phase: Participants will crossover to the intervention phase after 12 months. (Experimental): After a period of 12 months when all sites are in the control phase, crossover into the intervention phase will begin. The multilevel intervention will be the HDP Implementation Bundle. Patient education will be provided at time of participants' enrollment. This will cover knowledge of normal BP parameters, complications of HDP, warning symptoms, and advice on appropriate measures to take. A free automated BP monitor (e.g., Omron Series 3) will be provided and patients will be trained on BP measurement and instructed to report daily BP recordings via text messaging (similar to our feasibility study). Additionally, there will be a standardized follow-up interval (determined by Aim 1 results) for all patients with HDP and provision of free antihypertensive medications, if needed.
  Interventions: Other: Hypertension Disorders of Pregnancy (HDP) Implementation Bundle

INTERVENTIONS:
Other: Hypertension Disorders of Pregnancy (HDP) Implementation Bundle — The HDP Implementation Bundle will consist of 4 main blocks namely; patient education, home BP monitoring, a contextualized follow-up protocol and provision of free anti-hypertensives if need. Collectively, these will lead to design and development of a contextualized home BP monitoring program.
  Arms: Intervention Phase: Participants will crossover to the intervention phase after 12 months.

SUMMARY:
The goal of this interventional study is to learn from patients and healthcare providers at 4 health institutions (study sites) in Abuja and Kano in Nigeria what ways to best develop the content of a Hypertensive Disorders of Pregnancy ( HDP) Management package for pregnant women, and evaluate the effectiveness of implementing this package in improving cardiovascular health of pregnant women. The main question it aims to answer is:

Will a contextualized home BP monitoring program lead to better BP control among patients with HDP in Nigeria?

DETAILED DESCRIPTION:
This study aims to contextualize, implement, and evaluate the feasibility, fidelity, and acceptability and effectiveness of: 1) postpartum remote blood pressure monitoring, 2) patient education, 3) development of a standardized postpartum follow-up protocol, and 4) provision of free and/or subsidized antihypertensive medications for patients with HDP in University of Abuja, Murtala Muhammad Specialist Hospital, National Hospital, Abuja and Aminu Kano Teaching Hospital all in Nigeria. These components collectively make up a contextualized postpartum BP monitoring program called the HDP Implementation Bundle. The long-term objective is to implement a contextualized and acceptable evidence-based postpartum home BP monitoring program with supporting services and components, at 4 tertiary care institutions in Nigeria, to improve postpartum BP control in patients with HDP using a multilevel approach.

ELIGIBILITY:
Inclusion Criteria:

* Postpartum adults (>18 years)
* postpartum emancipated minors (in accordance with the Nigerian guidelines for young persons' participation in research and reproductive health services)
* with diagnosis of HDP prior to delivery delivered at one of the participating sites able to provide informed consent.

Exclusion Criteria:

* unable to provide consent.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2025-06-02 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Between group difference in change in systolic BP from baseline to 6-week follow-up | Baseline to 6 weeks
  The change in systolic BP from baseline to 6-week follow-up between the intervention and control group

SECONDARY OUTCOMES:
Between group differences in change in diastolic BP at 6 weeks follow-up and change in both systolic an diastolic BP at 12 weeks | Baseline to 6(and 12) weeks
  The change in diastolic BP from baseline to 6-week follow-up between the intervention and control groups.
Between group differences in systolic and diastolic BP at 12 weeks follow-up | Baseline to 12 weeks
  The change mean systolic and diastolic BPs 12 weeks follow-up between the intervention and control group

OTHER OUTCOMES:
Incidence of serious adverse events (eg dizziness) [Safety Outcomes] | Baseline to 6 months
  Safety outcomes include incidence of serious adverse events (eg dizziness) collected via surveys and patient charts at 6- weeks,12-weeks and 6-months postpartum
Number of eligible patient participants who utilized the HDP Implementation Bundle (Reach) | Baseline up to 57 months
  Number, age, socio-demographics of patients who were enrolled in the HDP Implementation Bundle.
Between-group difference in change in systolic BP from baseline to 6-week follow-up (Effectiveness) | Baseline up to 6 weeks
  Did the HDP Implementation Bundle impact effectiveness outcomes?
Number of clinical sites where the HDP Implementation Bundle was widely utilized (Adoption) | Baseline up to 57 months
  Records and surveys assessed to establish whether the HDP Implementation Bundle was widely utilized at clinical sites. Patient enrolment in HDP Bundle, where at least 1 home BP measurement is reported among total participants.
Number of clinical sites where the HDP Implementation Bundle was implemented as intended (Implementation) | Baseline up to 57 months
  Clinical site records and surveys assessed to evaluate whether the HDP Implementation Bundle was implemented as intended per the study protocol.
Number of clinical sites and patients that continue use of the HDP Implementation Bundle post completion. (Maintenance) | End of study at month 57 to 1 year post-completion
  Can the HDP Implementation Bundle be sustained? Continued use of the HDP Implementation Bundle or its components post-implementation.
Incidence of adverse events of special interest [Safety & Exploratory Outcomes] | Baseline to 6 months
  Exploratory outcomes include incidence of adverse events of special interest (e.g., dizziness, syncope, acute kidney injury) that will be collected via surveys and patient charts at 6- weeks,12-weeks and 6-months postpartum that could form the basis of new research questions or useful in developing hypotheses for exploring new research foci.
Between-group differences in change in diastolic BP at 6 weeks. (Effectiveness) | Baseline up to 6 weeks
  Did the HDP Implementation Bundle impact effectiveness outcomes
Between-group differences in change in systolic BP at 12 weeks. (Effectiveness) | Baseline to 12 weeks
  Did the HDP Bundle impact effectiveness outcomes?
Between-group differences in change in diastolic BP at 12 weeks. (Effectiveness) | Baseline to 12 weeks
  Did the HDP Implementation Bundle impact effectiveness outcomes?
Between-group differences in change in proportion of BP control at 6 weeks. (Effectiveness) | Baseline up to 6 weeks
  Did the HDP Implementation Bundle impact effectiveness outcomes
Between-group differences in change in proportion of BP control at 12 weeks. (Effectiveness) | Baseline to 12 weeks
  Did the HDP Implementation Bundle impact effectiveness outcomes?
Composite rate of fatal and nonfatal cardiovascular disease events. [Safety and Exploratory Outcomes] | Baseline up to 6 months
  The composite rate of fatal and nonfatal cardiovascular disease events will be calculated as the total sum of both fatal and nonfatal events out of the total study population times a hundred at 6 weeks, 12 weeks and 6 months as follows:
  Composite CVD Event Rate= (Total Study Population/Total Fatal + Nonfatal Events) ×100

CONTACTS AND LOCATIONS:
Overall Officials: Zainab Mahmoud, MD, MSc, Principal Investigator — Washington University School of Medicine
Locations (4):
- Nigeria (4):
  - National Hospital, Abuja, Abuja
  - University of Abuja Teaching Hospital, Abuja
  - Aminu Kano Teaching Hospital, Kano
  - Murtala Muhammad Specialist Hospital, Kano

IPD SHARING:
Plan to Share IPD: Yes
All data will be securely captured and stored within the University of Abuja REDCap system. The investigators will seek IRB approval from Washington University in St. Louis to access and analyze potentially identifiable information for the proposes of data analysis across the study aims. Data will be stored in secure, password protected servers with audit trails and accessibility only to trained study team members who have received IRB approval for access. The investigators will comply with the NIH policy for Data Management and Sharing (NOT-OD-21-013) and will share our protocol, data dictionary, statistical code and analysis plan with others, as soon as possible, and no later than time of an associated publication or end of the award period, whichever comes first.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: April 2029 - April 2034
Access Criteria: Access to this data will be made available via BioLINCC in accordance with NHLBI guidelines and due process, as this will be a controlled access database. All individuals requesting the data must submit an application with a research plan and documentation of review by an IRB.

REFERENCES:
- [Background] Federal Ministry of Health. Nigeria hypertension treatment protocol for the primary care level. Available at: https://linkscommunity.org/assets/PDFs/nigeria-hypertension-protocol-04.pdf.
- [Background] Petersen EE, Davis NL, Goodman D, Cox S, Syverson C, Seed K, Shapiro-Mendoza C, Callaghan WM, Barfield W. Racial/Ethnic Disparities in Pregnancy-Related Deaths - United States, 2007-2016. MMWR Morb Mortal Wkly Rep. 2019 Sep 6;68(35):762-765. doi: 10.15585/mmwr.mm6835a3. PMID 31487273
- [Background] Petersen EE, Davis NL, Goodman D, Cox S, Mayes N, Johnston E, Syverson C, Seed K, Shapiro-Mendoza CK, Callaghan WM, Barfield W. Vital Signs: Pregnancy-Related Deaths, United States, 2011-2015, and Strategies for Prevention, 13 States, 2013-2017. MMWR Morb Mortal Wkly Rep. 2019 May 10;68(18):423-429. doi: 10.15585/mmwr.mm6818e1. PMID 31071074
- [Background] Mahmoud Z, Joynt Maddox KE, Deych E, Lindley KJ. Racial Disparities in Specific Maternal Cardiovascular Outcomes. Circ Cardiovasc Qual Outcomes. 2022 Dec;15(12):e009529. doi: 10.1161/CIRCOUTCOMES.122.009529. Epub 2022 Nov 28. No abstract available. PMID 36440578
- [Background] Howell EA. Reducing Disparities in Severe Maternal Morbidity and Mortality. Clin Obstet Gynecol. 2018 Jun;61(2):387-399. doi: 10.1097/GRF.0000000000000349. PMID 29346121
- [Background] Lindley KJ, Aggarwal NR, Briller JE, Davis MB, Douglass P, Epps KC, Fleg JL, Hayes S, Itchhaporia D, Mahmoud Z, Moraes De Oliveira GM, Ogunniyi MO, Quesada O, Russo AM, Sharma J, Wood MJ; American College of Cardiology Cardiovascular Disease in Women Committee and the American College of Cardiology Health Equity Taskforce. Socioeconomic Determinants of Health and Cardiovascular Outcomes in Women: JACC Review Topic of the Week. J Am Coll Cardiol. 2021 Nov 9;78(19):1919-1929. doi: 10.1016/j.jacc.2021.09.011. PMID 34736568
- [Background] Ogunniyi MO, Mahmoud Z, Commodore-Mensah Y, Fleg JL, Fatade YA, Quesada O, Aggarwal NR, Mattina DJ, Moraes De Oliveira GM, Lindley KJ, Ovbiagele B, Roswell RO, Douglass PL, Itchhaporia D, Hayes SN; American College of Cardiology Cardiovascular Disease in Women Committee and the American College of Cardiology Health Equity Taskforce. Eliminating Disparities in Cardiovascular Disease for Black Women: JACC Review Topic of the Week. J Am Coll Cardiol. 2022 Nov 1;80(18):1762-1771. doi: 10.1016/j.jacc.2022.08.769. PMID 36302590
- [Background] WHO Recommendations for Prevention and Treatment of Pre-Eclampsia and Eclampsia - NCBI Bookshelf. https://www.ncbi.nlm.nih.gov/books/NBK140561/. Accessed 7 Feb 2023
- [Background] Bond RM, Gaither K, Nasser SA, Albert MA, Ferdinand KC, Njoroge JN, Parapid B, Hayes SN, Pegus C, Sogade B, Grodzinsky A, Watson KE, McCullough CA, Ofili E; Association of Black Cardiologists. Working Agenda for Black Mothers: A Position Paper From the Association of Black Cardiologists on Solutions to Improving Black Maternal Health. Circ Cardiovasc Qual Outcomes. 2021 Feb;14(2):e007643. doi: 10.1161/CIRCOUTCOMES.120.007643. Epub 2021 Feb 10. PMID 33563007
- [Background] United Nations Sustainable Development Goals. https://www.un.org/sustainabledevelopment/health/. Accessed 8 May 2023
- [Background] Charting the Future Together: The NHLBI Strategic Vision. https://www.nhlbi.nih.gov/sites/default/files/2017-11/NHLBI-Strategic-Vision-2016_FF.pdf. Accessed 15 May 2023
- [Background] Garovic VD, Dechend R, Easterling T, Karumanchi SA, McMurtry Baird S, Magee LA, Rana S, Vermunt JV, August P; American Heart Association Council on Hypertension; Council on the Kidney in Cardiovascular Disease, Kidney in Heart Disease Science Committee; Council on Arteriosclerosis, Thrombosis and Vascular Biology; Council on Lifestyle and Cardiometabolic Health; Council on Peripheral Vascular Disease; and Stroke Council. Hypertension in Pregnancy: Diagnosis, Blood Pressure Goals, and Pharmacotherapy: A Scientific Statement From the American Heart Association. Hypertension. 2022 Feb;79(2):e21-e41. doi: 10.1161/HYP.0000000000000208. Epub 2021 Dec 15. PMID 34905954
- [Background] Tukur J, Lavin T, Adanikin A, Abdussalam M, Bankole K, Ekott MI, Godwin A, Ibrahim HA, Ikechukwu O, Kadas SA, Nwokeji-Onwe L, Nzeribe E, Ogunkunle TO, Oyeneyin L, Tunau KA, Bello M, Aminu I, Ezekwe B, Aboyeji P, Adesina OA, Chama C, Etuk S, Galadanci H, Ikechebelu J, Oladapo OT; Maternal and Perinatal Database for Quality, Equity and Dignity Network. Quality and outcomes of maternal and perinatal care for 76,563 pregnancies reported in a nationwide network of Nigerian referral-level hospitals. EClinicalMedicine. 2022 Apr 28;47:101411. doi: 10.1016/j.eclinm.2022.101411. eCollection 2022 May. PMID 35518118
- [Background] Alliance for Maternal and Newborn Health Improvement (AMANHI) mortality study group. Population-based rates, timing, and causes of maternal deaths, stillbirths, and neonatal deaths in south Asia and sub-Saharan Africa: a multi-country prospective cohort study. Lancet Glob Health. 2018 Dec;6(12):e1297-e1308. doi: 10.1016/S2214-109X(18)30385-1. Epub 2018 Oct 22. PMID 30361107
- [Background] Trends in maternal mortality 2000 to 2020: estimates by WHO, UNICEF, UNFPA, World Bank Group and UNDESA/Population Division. https://www.who.int/publications/i/item/9789240068759.